CLINICAL TRIAL: NCT00567346
Title: A Randomised, DB, Plcb Controlled, Multicentre, Multinational Phase II/III Study to Assess the Efficacy and Safety of Three Different Dose Regimens of Oralgen Grass Pollen in Patients With Grass Pollen Related Allergic Rhinoconjunctivitis
Brief Title: Efficacy and Safety of Grass Pollen Sublingual Immunotherapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Artu Biologicals (Industry)
Responsible Party: Dr. F.F. Roosien, Artu Biologicals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AB0602; 2006-001548-30 (EudraCT Number)
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: randomised; double-blind; placebo-controlled; efficacy and safety; Oralgen® Grass Pollen; allergic rhinoconjunctivitis; Allergy; Rhinoconjunctivitis; Immunotherapy; Grass pollen extract
MeSH Terms: conditions — Hypersensitivity | interventions — grass pollen extract, alum-adsorbed

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- grass pollen extract twice weekly (Active Comparator): Current standard dose regimen of grass pollen immunotherapy (9,500 BU), given twice weekly. Note: patients in twice weekly dosing regimen will also receive placebo on days no active treatment is given.
  Interventions: Drug: Oralgen
- Grass pollen extract, daily (Active Comparator): Grass pollen immunotherapy, 9,500 BU, given daily
  Interventions: Drug: Oralgen
- Increased dose of grass pollen extract (Active Comparator): Increased dose of grass pollen immunotherapy, 19,000 BU, given daily
  Interventions: Drug: Oralgen
- Placebo control (Placebo Comparator): Patients randomized to placebo will receive placebo daily.
  Interventions: Drug: grass pollen extract

INTERVENTIONS:
Drug: Oralgen — Patients will receive drops of grass pollen immunotherapy sublingually
  Other Names: grass pollen extract
  Arms: Grass pollen extract, daily; Increased dose of grass pollen extract; grass pollen extract twice weekly
Drug: grass pollen extract — Patients will receive matching placebo sublingually
  Other Names: Placebo control
  Arms: Placebo control

SUMMARY:
The study is assessing efficacy and safety of three different dosage regimens of grass pollen sublingual immunotherapy in adult patients suffering from grass pollen related rhinoconjunctivitis.

DETAILED DESCRIPTION:
Patients with seasonal grass pollen related rhinoconjunctivitis will be randomized to one of four treatment groups at 41 centres in Europe. Each treatment group will consist of approximately 150 patients and 150 patients will be randomized to a placebo group. The study will consist of a screening phase, a treatment phase and a variable maintenance period.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 18-50
* patients with grass pollen related allergic rhinoconjunctivitis for at least 2 pollen seasons
* Positive skin prick test and IgE value of at least Class 2+
* RTSS of greater or equal to 14 during pollen season prior tot the start of the study
* Patients must be in general good health
* Patients with normal spirometry
* Informed consent given and willing to comply with the protocol
* Female patients are eligible if they use an accepted contraceptive method
* Negative urine pregnancy test if female

Exclusion Criteria:

* Pregnancy, breast feeding
* Asthma requiring treatment other than beta-2 inhaled agonists
* patients who have taken oral steroids within 12 weeks before screening visit
* patients who have received desensitisation treatment for grass pollen
* treatment by immunotherapy with any other allergen within the previous 5 years
* patients who have suffered a lower respiratory tract infection within 4 weeks or an upper respiratory tract infection within 2 weeks of the screening visit
* patients at risk of non-compliance
* participation in any other clinical study within the previous 3 months
* patients with a past or current disease, which may affect participation in or outcome of this study.
* patients treated with beta-blockers or under continuous corticotherapy
* allergic sensitivity to epithelial allergens the patients is exposed to
* positive skin prick test for environmental allergens and suffering from serious allergic symptoms due to exposure to these allergens during study period
* intention to subject the patient to surgery of the nasal cavity during current study
* Usual contraindications of immunotherapy
* a clinical history of symptomatic seasonal allergic rhinitis and/or asthma due to tree pollen or weed pollen adjacent to the start of, and potentially overlapping the grass pollen season

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 605 (Actual)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Primary efficacy variable is based on pollen season rhinoconjunctivitis Total Symptom Score (PS.RTSS) | One year

SECONDARY OUTCOMES:
Diarised Period RTSS on severity of rhinoconjunctivitis scores and rescue medication usage will be calculated to assess efficacy. Safety will be assessed through AE profile, the assessment of routine safety tests. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Folkert R Roossien, Study Director — Artu-Biologicals Europe B.V., the Netherlands
Locations (40):
- Bulgaria (6):
  - MHAT PLovdiv, ENT Clinic, Plovdiv
  - 5th MHAT, ENT Clinic, Sofia
  - Military Medical Academy, Sofia
  - Ministry of interior-central clinical database, Sofia
  - MHAT Sveta Marina, Varna
  - Military Medical Academy, Varna
- Czechia (9):
  - ORL Soukroma praxe, Brno
  - Fakultni nemocnice Brno, Brno-Bohunice
  - Nemocnice Caslav, Čáslav
  - Alergologicka ordinace, Dobruška
  - Alergologicka ambulance, Jablonec nad Nisou
  - Alergologicka ordinace, Kutná Hora
  - Alergologicka ambulance, Ostrava - Hrabuvka
  - Ambulance plicni a alergologicka, Ostrave - Hrabuvka
  - Alergologicka ambulance Okresni nemocnice Tabor, Tábor
- Germany (6):
  - Berufsgen. kliniken Bergmannsheil, Bochum
  - Univ. klinikum Carl Gustav Carus, Dresden
  - MedicoKIT, Goch
  - Johannes-Gutenberg-Universitat Mainz, Mainz
  - Vital Care, München
  - Privataertz. inst. & Forsh. einrichtung, Wiesbaden
- Hungary (5):
  - Svabhegyi Allami Gyermekgyogyintezet pulmonologia, Budapest
  - Szent Janos Korhaz, Budapest
  - Selye Janos Korhaz, Komárom
  - Karolina Korhaz, Mosomagyarovar
  - Tudogyogyintezet Torokbalint, Törökbálint
- Lithuania (5):
  - Kaunas medical University hospital, Kaunas
  - Klaipeda Regional Hospital, Klaipėda
  - JSC Seimos gydytojas, Vilnius
  - Vilnius Central Outpatient Clinic, Vilnius
  - Vilnius university hospital, Santariskiu Clinic, Vilnius
- Netherlands (4):
  - Ampha, 's-Hertogenbosch
  - Ampha, De Bilt
  - Ampha, Hengelo
  - Menox, Nijmegen
- Slovakia (5):
  - Centrum imunologie a alergologie s.r.o, Bratislava
  - FNsP Nove Zamky, ambulancia TaRCh, Nové Zámky
  - Amb. klinickey imunologie a allergologie UTaRCH, Poprad
  - Ambulancia klinickej imunologie a alergologie, Trenčín
  - Medcentrum s.r.o., Žilina